CLINICAL TRIAL: NCT02190448
Title: A Randomized, Placebo-Controlled Study of an Herbal Tea to Support Lactation
Brief Title: Randomized, Placebo-Controlled Study of an Herbal Tea to Support Lactation
Acronym: SLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Traditional Medicinals Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SLS2013
Record Dates: First submitted 2013-07-15; First posted 2014-07-15 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Lactation
Keywords: galactogogue; lactation; milk production; breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study herbal tea (Experimental): Supplementation of 3-5, 8 oz cups of study tea daily for 4 weeks.
  Interventions: Dietary Supplement: study herbal tea
- herbal placebo tea (Placebo Comparator): Supplementation of 3-5, 8oz cups of tea daily for 4 weeks.
  Interventions: Dietary Supplement: herbal placebo tea

INTERVENTIONS:
Dietary Supplement: study herbal tea — 3-5 cups, 8oz tea daily for 4 weeks
  Arms: study herbal tea
Dietary Supplement: herbal placebo tea — 3-5 cups, 8oz each daily for 4 weeks
  Arms: herbal placebo tea

SUMMARY:
The overall aims of this project are to 1) determine the quality of life effects of a combination herbal galactagogue tea in lactating women, and 2) measure changes in maternal blood concentration of oxytocin, prolactin, and milk production. The defined outcome measures will include quality of life measures in the breastfeeding woman and basic infant health. If the tea proves safe and effective, then it can provide a proven all-natural and organic supplement for increasing lactation in women. This in turn will increase quality of life for both the infant and the mother.

DETAILED DESCRIPTION:
In order to establish the quality of life of combination herbal galactagogue tea in lactating women, a randomized controlled trial of combination herbal galactagogue tea vs. placebo is being undertaken in 120 fully lactating women beginning at 2-12 weeks postpartum for four weeks. Women will be randomized to one of two teas: combination herbal galactagogue tea vs. an herbal placebo tea. The study duration will be 4 weeks total beginning in the second to twelfth week postpartum, with follow up phone calls at postpartum months 3, 6, 9 and 12, to ascertain if the mother is continuing to breastfeed. During the 4-week study, participants and their infants will have three scheduled outpatient visits to the Medical University of South Carolina or an affiliated study center: one visit at 2-12 weeks postpartum, a second visit at 4-14 weeks postpartum, and a final visit at 6-16 weeks postpartum. The first visit, will include watching a video on how to correctly steep the tea and then brewing tea in the presence of the study coordinator, in addition to the procedures listed below. This initial visit will last approximately 90 minutes. Each subsequent visit will take less than 60 minutes for a maternal blood drawing, pumping a breast milk sample, answering questionnaires, and both weighing and measuring the infant. Study participants will be given a study journal to be completed with the number of cups of tea they drink every day and to document an assessment of how they felt throughout the day both physically and emotionally. All participants will receive telephone calls/texts, depending on the study participants preferred method of communication. This will be done by a Study Coordinator at the end of weeks 1 and 3 of the study in order to ensure safety and to remind them to complete their journals. This call will also be an opportunity to assess if the participant is in need of additional dietetic or lactation support by the team professionals or if she is having any difficulty brewing her tea. At the last study visit, participants will be asked to call and report any adverse events for 3 months after the end of their time on the active study.

Post Active-Study Communication: After the active-study, the Study Coordinators will call each study participant when their infants are 3, 6, 9 and 12 months old, if applicable in order to record the number of months that she continues to fully or partially breastfeed.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 45 years
* Good general health
* Lactating
* Singleton birth
* Two to twelve weeks postpartum
* Have a full term (>37 weeks gestation) healthy infant
* Is successfully fully breastfeeding at the time they enter the study
* Intend to fully breastfeed their infants for the following 4 weeks at the time of enrollment.

Exclusion Criteria:

* Chronic illnesses (e.g. diabetes, hypertension, bronchial asthma, Gastroesophageal Reflux Disease (GERD), atopic dermatitis, celiac disease or gluten sensitivity, Crohn's Disease, ulcerative colitis, eating disorders, breast cancer, blood disorder, psychiatric)
* Pre-pregnant BMI (>50)
* History of alcohol, drug abuse or cigarette smoking
* Currently using the following pharmaceuticals: diuretics, pseudoephedrine, anticholinergics, and an estrogen-containing birth control pill or using an estrogen-containing device
* Currently consuming other drugs/herbals used to induce milk production including metoclopramide, domperidone, or other drugs/herbals (i.e. fenugreek capsules, goat's rue products, or "More Milk" capsules or tinctures)
* Sensitivity or known allergies to peanuts, soybeans, or chick peas
* Sensitivity or known allergies to plants in the Apiaceae/carrot plant family (e.g. anise, celery, coriander, fennel) or the compound anethole
* Sensitivity or known allergies to plants in the Asteraceae/daisy family (e.g. blessed thistle, echinacea, or calendula)
* Taking a selective serotonin reuptake inhibitor (SSRI)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Quality of life | 4 weeks
  To determine quality of life, the following measurement tools will be compared across the 3 study visits:
  • The Satisfaction with Life Scale (Diener, Emmons et al. 1985; Pavot, Diener et al. 1991; Pavot and Diener 1993; Shevlin, Brunsden et al. 1998)-an overall global life satisfaction questionnaire.
Quality of life | 4 weeks
  To determine quality of life, the following measurement tools will be compared across the 3 study visits:
  • World Health Organization's World Health Organization Quality of Life - Brief Survey [WHOQOL-BREF] (WHO 1997; Skevington, Lotfy et al. 2004)-Current perception of position in life in context of personal culture and value systems.
Quality of life | 4 weeks
  To determine quality of life, the following measurement tools will be compared across the 3 study visits:
  • Edinburgh Postpartum Depression Inventory:(Murray and Carothers 1990)-a postpartum depression screen
Quality of life | 4 weeks
  To determine quality of life, the following measurement tools will be compared across the 3 study visits:
  • State-Trait Anxiety Inventory (STAI-Y) (Spielberger, Gorsuch et al. 1970; Ramanaiah, Franzen et al. 1983; Spielberger and Vagg 1984) -differentiates between temporary or emotional state anxiety versus long standing personality trait anxiety in adults.

SECONDARY OUTCOMES:
Oxytocin in maternal blood | 4 weeks
  Blood will be collected at each of the 3 study visits. We will measure changes in maternal blood concentrations of oxytocin, across study groups.
Prolactin in maternal blood | 4 weeks
  Blood will be collected at each of the 3 study visits. We will measure changes in maternal blood concentrations of prolactin, across study groups.
Composition of breast milk | 4 weeks
  Measuring the quantities and quality of breast milk at the 3 study visits between groups. Checking the composition for milk caloric density and fatty acid content between the placebo and the combination galactagogue tea.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Marriott, PhD, Principal Investigator — Medical University of South Carolina; Carol Wagner, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Academy Of Breastfeeding Medicine Protocol Committee. ABM Clinical Protocol #9: Use of galactogogues in initiating or augmenting the rate of maternal milk secretion (First Revision January 2011). Breastfeed Med. 2011 Feb;6(1):41-9. doi: 10.1089/bfm.2011.9998. PMID 21332371
- [Background] Turkyilmaz C, Onal E, Hirfanoglu IM, Turan O, Koc E, Ergenekon E, Atalay Y. The effect of galactagogue herbal tea on breast milk production and short-term catch-up of birth weight in the first week of life. J Altern Complement Med. 2011 Feb;17(2):139-42. doi: 10.1089/acm.2010.0090. Epub 2011 Jan 24. PMID 21261516
- [Derived] Foong SC, Tan ML, Foong WC, Marasco LA, Ho JJ, Ong JH. Oral galactagogues (natural therapies or drugs) for increasing breast milk production in mothers of non-hospitalised term infants. Cochrane Database Syst Rev. 2020 May 18;5(5):CD011505. doi: 10.1002/14651858.CD011505.pub2. PMID 32421208
- See also: Steeped with Love Study — https://www.facebook.com/SteepedwithLoveStudy